CLINICAL TRIAL: NCT05842174
Title: Targeting Ischemia-Induced Autophagy Dependence in Hepatocellular Carcinoma Through Image-guided Locoregional Therapy
Brief Title: Targeting Ischemia-Induced Autophagy Dependence in Hepatocellular Carcinoma
Acronym: TAQE
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ONCC-008-22S; IO1CX002542 (Other Grant/Funding Number: VA CSR&D)
Record Dates: First submitted 2023-04-05; First posted 2023-05-03 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular carcinoma; Transarterial Chemoembolization; Transarterial Embolization; Autophagy
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Hydroxychloroquine; Ethiodized Oil

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Transarterial Embolization with Hydroxychloroquine (Experimental): Intra-arterial hydroxychloroquine in Lipiodol + transarterial embolization followed by oral hydroxychloroquine
  Interventions: Drug: Hydroxychloroquine; Drug: Lipiodol
- Transarterial Embolization without Hydroxychloquine (Placebo Comparator): Intra-arterial Lipiodol + transarterial embolization followed by oral placebo
  Interventions: Drug: Lipiodol; Drug: Placebo

INTERVENTIONS:
Drug: Hydroxychloroquine — Hydroxychloroquine to be administered intra-arterially at time of transarterial embolization as well as orally for 6 weeks following the procedure
  Arms: Transarterial Embolization with Hydroxychloroquine
Drug: Lipiodol — Lipiodol is an FDA-approved drug delivered agent and embolic which is administered as standard of care for transarterial embolization for hepatocellular carcinoma. Lipiodol will be administered intra-arterially in both arms at the time of procedure.
Drug: Placebo — Placebo will be administered orally for 6 weeks following the procedure to patients in arm 2
  Arms: Transarterial Embolization without Hydroxychloquine

SUMMARY:
Trans-arterial chemoembolization (TACE) is the most commonly used therapy for patients with unresectable hepatocellular carcinoma (HCC). TACE is a minimally invasive procedure that involves placing a catheter into the artery in the liver that feeds the tumor, administering chemotherapeutics and then blocking the artery with embolics in order to kill tumor cells by depriving them of essential oxygen and nutrients. While TACE has a proven survival benefit, local recurrence is common, and long-term survival rates are poor. Prior studies demonstrate that HCC cells survive the oxygen and nutrient deprivation through autophagy, a process of cellular self-eating, to provide nutrients required for survival. The proposed project will leverage this dependency to develop a novel approach to TACE that integrates autophagy inhibition to improve therapeutic response by increasing tumor cell killing and enhancing anti-tumor immunity.

DETAILED DESCRIPTION:
Surgical resection or liver transplantation remain the only curative options for patients with hepatocellular carcinoma (HCC). However, fewer than 20% of patients with HCC are candidates for resection. Transarterial embolization with or without chemotherapy (TA(C)E) is an endovascular locoregional embolotherapy that involves hepatic artery embolization with intra-arterial infusion of a chemotherapeutic agent. TA(C)E is considered the standard of care for treating unresectable HCC in the remaining 80% of patients. While TA(C)E has a proven survival benefit, local recurrence is common, and long-term survival rates are poor. Moreover, only 44% of treated HCCs demonstrate extensive necrosis on pathology following TA(C)E, indicating tumor cells develop an adaptive metabolic stress response (MSR) enabling their survival under TA(C)E-induced nutrient and oxygen deprivation.

In preliminary studies, the investigators have demonstrated that HCC cells are pre-programmed to survive TA(C)E-induced ischemia through enhanced function of autophagy. Moreover, TA(C)E-induced ischemia results in quiescence in surviving HCC cells and a dependence on autophagy. As such, these data demonstrate that TA(C)E offers a unique opportunity to constrain metabolic phenotypes in order to generate this targetable dependency in HCC. The proposed project will build on this prior work to: 1) study a novel TA(C)E paradigm which targets this ischemia-induced dependency on autophagy using hydroxychloroquine (HCQ) and 2) characterizes the efficacy and evolution of autophagy inhibition using HCQ as well as associated alterations in anti-tumor immunity. To achieve these goals, this submission proposes a first in human, early phase prospective clinical trial to assess the safety and efficacy of autophagy inhibition using intra-arterial (IA) HCQ with TAE followed by maintenance of autophagy inhibition with daily oral HCQ for 6 weeks following embolization. Follow-up tumor biopsies and serum sampling 3-4 and 5-6 weeks after embolization will inform on the on-target efficacy of autophagy inhibition and its effect on the tumor microenvironment and immune response.

This trial will pursue three aims: (1) to establish the clinical safety of the combination of the autophagy inhibitor HCQ with TAE to treat patients with intermediate stage HCC (phase 1); (2) to compare the short-term efficacy of HCQ with TAE versus TAE alone in patients with intermediate stage HCC (phase 2); and (3) to characterize differences in local and systemic immune modulation following TAE as compared to IA HCQ TAE.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18 years, meeting criteria for diagnosis of BCLC B HCC and referred to undergo TACE
* HCC measuring 3 cm in minimum transverse diameter and meets LI-RADS 5 criteria based on cross-sectional imaging as determined by a board-certified, sub-specialty trained radiologist
* Childs Pugh Turcotte A/B7, Performance Status 0
* Informed of investigational nature of this study with provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study

Exclusion Criteria:

* QT prolongation on ECG
* Retinopathy on ophthalmologic examination
* Females who are pregnant or breast feeding at the time of screening will not be eligible for this study

  * a serum or urine pregnancy test will be performed in women of child-bearing potential at screening
* Prior LRT or systemic therapy to the target lesion
* Contraindication to contrast enhanced MRI or metallic implant within the liver.
* HCQ allergy, porphyria, uncontrolled psoriasis, and existing retinopathy
* Lesion not amenable to biopsy based on pre-TACE imaging as determined by treating interventional radiologist
* Serious or unstable medical or psychological conditions that, in the opinion of the investigator, would compromise the subject's safety or successful participation in the study)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2029-09-30 (Estimated); Study Completion 2030-10-15 (Estimated)

PRIMARY OUTCOMES:
Local Progression Free Survival | 6 months following treatment
  Local progression free survival will be determined on a per lesion basis based on follow-up cross-sectional imaging and modified response evaluation criteria in solid tumors

CONTACTS AND LOCATIONS:
Overall Officials: Terence P Gade, MD PhD, Principal Investigator — Corporal Michael J. Crescenz VA Medical Center, Philadelphia, PA
Locations (1):
- Corporal Michael J. Crescenz VA Medical Center, Philadelphia, PA, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No